CLINICAL TRIAL: NCT01058317
Title: Propranolol Administration in Pediatric Patients With Recurrent Respiratory Papillomatosis
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: No participants enrolled
Sponsor: Massachusetts Eye and Ear Infirmary (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-10-104
Record Dates: First submitted 2010-01-27; First posted 2010-01-28 (Estimated); Last update posted 2013-11-21 (Estimated); Status verified 2012-04

CONDITIONS: Recurrent Respiratory Papillomatosis
Keywords: respiratory, papilloma, pediatric, juvenile
MeSH Terms: conditions — Recurrent respiratory papillomatosis; Papilloma | interventions — Propranolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Children treated with propranolol (Experimental)
  Interventions: Drug: Propranolol

INTERVENTIONS:
Drug: Propranolol — Propranolol 2mg/kg divided twice daily

SUMMARY:
Juvenile onset recurrent respiratory papillomatosis (JORRP) is a rare, difficult to treat, benign tumor of the pediatric airway. Current therapy is mainly surgical, but in a significant portion of patients adjuvant therapy is required to control the disease process. Although multiple adjuvant medical therapies have been tried, success has been limited. We have seen some success in a limited amount of patients using orally administered propranolol. Our goal is to enroll a larger cohort of patients to determine the effectiveness of propranolol as an adjuvant therapy for JORRP.

ELIGIBILITY:
Inclusion Criteria:

* 1. Biopsy proven with appropriate Human Papilloma Virus typing Recurrent Respiratory Papilloma
* 2. Child under age 10
* 3. Informed consent and where appropriate informed assent
* 4. Children who have undergone at least 4 documented surgical interventions in the past year.

Exclusion Criteria:

* Parental or child refusal to participate
* Heart failure
* Atrio-ventricular heart block
* Cardiac anomalies
* Low resting heart rate
* Low resting blood pressure
* Wolff-Parkinson White Syndrome
* Unexplained syncope
* Asthma or Reactive airway disease
* Renal or liver failure
* Expected long fasting periods, >12 hours
* Diabetes Mellitus
* Hypersensitivity to propranolol

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2010-01; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Decreased number of surgeries | 3 months

SECONDARY OUTCOMES:
Improved voice quality | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Hartnick, MD, Principal Investigator — Massachusetts Eye and Ear Infirmary